CLINICAL TRIAL: NCT06339151
Title: Efficacy of Intravenous Dexamethasone Injection Given 12 and 24 Hours for Pain After Total Knee Arthroplasty: A Prospective Randomized Clinical Trial
Brief Title: Comparing Single Dose and Multiple Dose of Dexamethasone Post TKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Dr., Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUH multiple dexamethasone TKA
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-04

CONDITIONS: Osteo Arthritis Knee; Pain, Postoperative
Keywords: total knee arthroplasty; dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Preoperative - Dexamethasone 0.15 mg/kg injection by the anesthesiologist 30 minutes before surgery.
  Postoperative 12 hr - Normal saline solution injection Postoperative 24 hr - Normal saline solution injection
  Interventions: Drug: Dexamethasone before surgery
- Group 2 (Active Comparator): Preoperative - Dexamethasone 0.15 mg/kg injection by the anesthesiologist 30 minutes before surgery.
  Postoperative 12 hr - Dexamethasone 0.15 mg/kg IV at 12 hours post operation Postoperative 24 hr - Normal saline solution injection
  Interventions: Drug: Dexamethasone before and 12 hours after surgery
- Group 3 (Active Comparator): Preoperative - Dexamethasone 0.15 mg/kg injection by the anesthesiologist 30 minutes before surgery.
  Postoperative 12 hr - Normal saline solution injection Postoperative 24 hr - Dexamethasone 0.15 mg/kg IV at 24 hours post operation
  Interventions: Drug: Dexamethasone before and 24 hours after surgery

INTERVENTIONS:
Drug: Dexamethasone before surgery — Dexamethasone 0.15 mg/kg IV before surgery
  Arms: Group 1
Drug: Dexamethasone before and 12 hours after surgery — Dexamethasone 0.15 mg/kg IV before surgery Dexamethasone 0.15 mg/kg IV at 12 hours post operation
  Arms: Group 2
Drug: Dexamethasone before and 24 hours after surgery — Dexamethasone 0.15 mg/kg IV before surgery Dexamethasone 0.15 mg/kg IV at 24 hours post operation
  Arms: Group 3

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of single dose and double dose of dexamethasone after primary total knee replacement.

The main question[s] it aims to answer [is/are]:

Does 24 hours-interval of double dose of dexamethasone have better analgesic effect than single dose and 12 hours interval of double dose of dexamethasone after primary total joint replacement?

Researchers will compare double dose of dexamethasone group to see if [insert effects].

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
1. Randomized patients into 3 groups

   * Group 1: Patients received only Dexamethasone 0.15 mg/kg IV before surgery.
   * Group 2: Patients received Dexamethasone 0.15 mg/kg IV before surgery and Dexamethasone 0.15 mg/kg at 12 hours after surgery.
   * Group 3: Patients received Dexamethasone 0.15 mg/kg before surgery along and Dexamethasone 0.15 mg/kg at 24 hours after surgery.
2. Preemptive analgesia Alprazolam 0.5 mg. 1 tablet, Pregabalin 75 mg. 1 tablet before bedtime Celecoxib 400 mg. 1 tablet, Omeprazole 20 mg 1 mg tablet, Paracetamol 500 mg 2 tablets and 1 Ondansetron 4 mg 1 tablet at 1 hour before surgery.
3. The researcher will give an injection. Dexamethasone 0.15 mg/kg injection form together with Cefazolin 1 gm injection form by the anesthesiologist 30 minutes before surgery.
4. Spinal Anesthesia by an anesthesiologist before surgery The anesthetic component consists of 0.5% Bupivacaine 15 mg, which does not contain morphine, along with local anesthesia in the thigh area (Adductor canal block) with a mixture of 0.5% Bupivacaine 15 mg.
5. All patients will undergo knee replacement surgery in the same manner
6. Periarticular cocktail injection The drug contains Tranexamic acid 10 mg/kg, Morphine 5 mg, Adrenaline 0.5 mg, 5% Bupivacaine 200 mg (Marcaine 1 amp), Ketorolac 30 mg (1 amp) mixed with saline (Normal saline) until 75 ml of area is obtained. The injection site is placed around the knee joint and knee capsule.
7. After surgery, the patient will stay in the recovery room for 2 hours to take care of their symptoms.
8. Pain relievers after surgery include

   * Parecoxib (Dynastat) 40 mg injection every 12 hours for the first 2 days after knee replacement surgery, then change the medicine to Celecoxib 400 mg. 1 tablet after breakfast
   * Paracetamol 500 mg. 2 tablets every 6 hours for the first 2 days after knee replacement surgery. After that, give Paracetamol 500 mg. 2 tablets pro for pain every 6 hours
   * Pregabalin 75 mg. 1 tablet po hs
   * Morphine 3 mg injection every 4 hours for patients with a pain score greater than 4 points (VAS-P score ≥4)
   * Ondansetron 4 mg IV prn for nausea and vomitting every 6 hours
   * Alprazolam 0.5 mg 1 tab po hs
   * Cefazolin 1 gm IV every 6 hours for the first 24 hours after surgery
9. Group 2 patients will receive Dexamethasone 0.15 mg/kg as an injection after surgery at 12 hours, and patients in Group 3 will receive Dexamethasone 0.15 mg/kg as injection at 24 hours after surgery

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis of knee joint
* Undergo unilateral primary total knee replacement
* Age between 50-85 years old

Exclusion Criteria:

* Allergy to dexamethasone
* History of long term corticosteroid used
* New York heart association (NYHA) class > II
* Type 2 Diabetes mellitus that had HbA1c > 7 % or FBS > 200 mg/dl
* Chronic kidney disease > stage III or eGFR < 60
* Cirrhosis Child class B or C
* Cannot use pain controlled as protocol
* History of previous knee surgery
* History of previous septic arthritis at knee joint

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain at rest and motion | At 6 hour, 12 hour, 18 hour, 24 hour, 30 hour, 36 hour, 42 hour, 48 hour, 54 hour, 60 hour, 66 hour and 72 hour after surgery
  Using visual analog scale 0-10 (0 means best, 10 means worst)

SECONDARY OUTCOMES:
Nausea and vomiting | At 24 hour, 48 hour and 72 hour after surgery
  Using visual analog scale 0-10 (0 means best, 10 means worst)
Morphine consumption | At 24 hour, 48 hour and 72 hour after surgery
  Total milligrams use of morphine postoperative (record in mg)
Blood sugar level | At 24 hour and 48 hour after surgery
  record in mg/dL
CRP level | At 24 hour and 48 hour after surgery
  record in mg/dL
Range of motion | At 24 hour and 48 hour after surgery
  Using long arm goniometer (record in degrees)
Length of hospital stay | up to 1 week
  Number of days the patient stays for surgery
Complication | up to 6 months
  Surgical site infection, deep infection or wound complication

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu H, Zhang S, Xie J, Lei Y, Cao G, Pei F. Multiple Doses of Perioperative Dexamethasone Further Improve Clinical Outcomes After Total Knee Arthroplasty: A Prospective, Randomized, Controlled Study. J Arthroplasty. 2018 Nov;33(11):3448-3454. doi: 10.1016/j.arth.2018.06.031. Epub 2018 Jul 4. PMID 30033064